CLINICAL TRIAL: NCT02988505
Title: Out-of Pocket Payments in Patients With Lymphedema in France and Inequities of Access ti Healthcare
Brief Title: Out-of Pocket Payments With Lymphedema in France
Acronym: Lymphorac
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF 9401
Record Dates: First submitted 2016-09-02; First posted 2016-12-09 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2016-08

CONDITIONS: Primary Lymphedema Secondary Lymphedema
MeSH Terms: interventions — Standard of Care; Pharmaceutical Preparations; Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Standard care
  Other Names: Standard care including medical visits , drugs and medical devices

SUMMARY:
Lymphedema is a frequent and chronic condition posing a high burden on patients. Clinical guidelines emphasize the role of compression therapy by prescription medical devices. Even in a mandatory publicly funded health insurance system, out-of-pocket payments (OOPP) may exist due to the price and reimbursement setting processes. OOPP may threaten the equity of care and drive patients to forgo care. Our aim was to analyze the distributive effects of OOPP for lymphedema patients in France.

A prospective, multicenter study will be conducted in France in 2014 on patients with lymphedema. Household ability to pay will be specified by net income and OOPP will be assessed prospectively over 6 months for outpatient care (visits, drugs, medical devices, nursing care, biological tests, imaging, physiotherapy and transportations). Both mandatory and voluntary health insurance reimbursements will be considered. We will combine concentration curves and concentration indices to assess the distributive effects.

ELIGIBILITY:
Inclusion criteria:

* Patient aged over six years, with primary or secondary lymphedema, regardless of the severity of the disease;
* Patient treated in one of the centres participating in the study;
* Patient (and her legal representative for minors) who gave her written consent [or did not refuse to participate, according to local Law] ;
* Patient with Internet access and an active email address.

Exclusion criteria:

* Patients with concomitant chronic venous insufficiency;
* Patient not covered by any health care insurance scheme;
* People protected under the law.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients meeting the inclusion criteria will be included in each participating centre during the inclusion phase
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The mean monthly out-of-pocket payment as assessed by an online self-questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Departement information Medicale CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No